CLINICAL TRIAL: NCT06180135
Title: The Effect Of Coffee And Tea Drink On Gis Functions Healing Quality After Surgery In Patients Surgery
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Eastern Mediterranean University (Other)
Responsible Party: Principal Investigator, Gülcan Dürüst Sakallı, lecturer, Eastern Mediterranean University
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: EasternMU-SBF-HB-GDS-02
Record Dates: First submitted 2023-07-26; First posted 2023-12-22 (Actual); Last update posted 2025-01-22 (Actual); Status verified 2025-01

CONDITIONS: Gastrointestinal Functions
Keywords: TURKİSH COFFE; FENNEL TEA; GIS FUNCTIONS; HEALING QUALITY; APAROSCOPIC CHOLECYSTECTOMY SURGERY

STUDY DESIGN:
Intervention Model Description: Therre Groups. Group were comprised of control group, fennel tea drink group, turkısh coffee drink group.
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (3):
- Control Group (No Intervention): The patients in this group will rest their bowel movements after starting oral intake at the 6th hour postoperatively. The time of first degassing and the time of first discharge will be recorded by asking verbally.
  Only evaluation will be made at 6. hours after surgery without intervention in the control group.
- TURKISH COFFEE DRINKING GROUP - TURKISH COFFEE DRINK (Active Comparator): Turkish coffee group after the patients in start oral intake at the 6th hour after the surgery, 7 gr of Turkish coffee in 75 ml of water will be boiled with water at 50-60°C, prepared by the researcher and given to the patients to drink. Bowel movements will be rested before and after the intake of Turkish coffee. The time of first degassing and the time of first discharge will be recorded by asking verbally.
  Evaluation will be made at the 0th hour after the operation without application. The application will be made at the 6th hour after the surgery and the gıs functıons and healıng qualıty will be evaluated.
  Interventions: Other: TURKISH COFFEE DRINK
- FENNEL TEA DRINKING GROUP- FENNEL TEA DRINK (Active Comparator): fennal tea group after the patients in start oral intake at the 6th hour postoperatively, 150 ml of boiled water at 100˚C will be added to 2 g of fennel seeds, and then infused for 5-10 minutes, they will be given to the patients to drink. Bowel movements will be rested before and after fennel tea intake. The time of first degassing and the time of first discharge will be recorded by asking verbally.
  Evaluation will be made at the 0th hour after the operation without application. The application will be made at the 6th hour after the surgery and the gıs functıons and healıng qualıty will be evaluated.
  Interventions: Other: FENNEL TEA DRINK

INTERVENTIONS:
Other: TURKISH COFFEE DRINK — TURKISH COFFEE DRINK
  Arms: TURKISH COFFEE DRINKING GROUP - TURKISH COFFEE DRINK
Other: FENNEL TEA DRINK — FENNEL TEA DRINK
  Arms: FENNEL TEA DRINKING GROUP- FENNEL TEA DRINK

SUMMARY:
The positive effects of coffee on general health, central nervous system, cardiovascular system and bowel movements in healthy people are known. In a few studies conducted in recent years, it is stated that coffee consumption is a safe and effective method for accelerating bowel movements after surgical intervention.

It is known that many plants have been used for medicinal purposes since ancient times in the world. Among these plants is fennel (foeniculum vulgare). The fennel plant was used as a spice in Greece and Rome, as well as recognized and used for medicinal purposes. Fennel, dyspeptic ailments; it is effective in spasmodic gastrointestinal complaints, bloating, gas and upper respiratory tract disorders This research; A randomized controlled study was planned to evaluate the effects of Turkish coffee and fennel tea consumption on patients' gastrointestinal functions and healing quality after laparoscopic cholecystectomy surgery.

DETAILED DESCRIPTION:
Surgical interventions can be large or small, planned or urgent, but they have physiological and psychological effects on people. The most obvious physiological effects on the patient are: deterioration of organ functions and vascular system, change in body image, activation of stress-alarm reaction. Another of these physiological effects and the most common one is the changes in the gastrointestinal system. Postoperative ileus, which is defined as the temporary deterioration of gastric motility, causes pre- and postoperative diet restrictions, administration of anesthetics/narcotics, delay in gastric emptying as a result of excessive use of isotonic solutions, and slowing down in bowel movements due to excessive touching of the intestines, especially in abdominal and pelvic surgeries. It is known that current approaches and evidence-based practices regarding treatment and care in surgery can accelerate post-surgical recovery and reduce surgery-related deaths. In this direction, one of the evidence-based applications that has emerged to accelerate post-operative recovery is Enhanced Recovery After Surgery - ERAS, also known as Fast Track Surgery (FTS) protocol. With these new approaches, it has been proven that the time between the onset of bowel movements and the first gas formation is shortened, wound healing is accelerated, infection rates are reduced, and hospital stay is reduced. One of these approaches is coffee consumption in the postoperative period. Coffee is a popular beverage and its effects on general health, the central nervous system and the cardiovascular system are well known. Caffeine is a moderate central nervous system stimulant, and these effects are mediated by adenosine receptors. It acts as a potential antagonist of adenosine receptors in the nervous system. Caffeine and adenosine molecules are similar molecules. Caffeine binds to adenosine receptors, thus reducing the effectiveness of adenosine. As a result, we feel the stimulating effect of caffeine at the highest level. It has been observed that consuming more than 7 cups of coffee per day increases gastric secretion. It is also known that coffee increases bowel movements in healthy people. In a study conducted with patients who underwent laparoscopic orectal surgery, it was determined that bowel movements started 3 hours earlier than the patients in the control group and stayed one day less in the hospital. However, in the literature review, it is observed that there are very limited studies on this subject.

In the literature review, early oral feeding, mobilization and gum chewing were found to be effective in preventing paralytic ileus after abdominal and laparoscopic surgery, increasing patient comfort and shortening hospital stay. However, studies examining the effect of coffee consumption on bowel movements and hospital stay in the early postoperative period are very limited.

Based on this information, this study was planned to evaluate the effects of Turkish coffee and fennel tea drinking on GIS functions and healing quality in patients who underwent laparoscopic laparoscopic cholecystectomy surgery.

ELIGIBILITY:
Inclusion Criteria:

* Patients who have undergone laparoscopic cholecystectomy under general anesthesia
* Patients whose bowel functions do not have all chronic or metabolic features,
* Patients without auditory, mental and past diseases
* Patients who volunteered for the study

Exclusion Criteria:

* Patients who did not receive general anesthesia and did not have laparoscopic cholecystectomy surgery
* Those who have any chronic or metabolic disease that will affect intestinal functions,
* Those with auditory, mental and neurological diseases,
* Patients using drugs for psychiatric disorders,
* who are not willing to participate in the research,
* Patients who are intubated and sedated,
* Those with stoma
* Patients with previous abdominal surgery will not be included in the study.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 108 (Actual)
Dates: Start 2023-08-05 (Actual); Primary Completion 2023-12-30 (Actual); Study Completion 2025-01-20 (Actual)

PRIMARY OUTCOMES:
Form For Evaluation Of The Patient's Gastrointestinal Functions | one day first 6 th hour
  Marking will be Yes or No. For example, is there gas output? yes/no
Quality Of Healing Scale | one day first 6 th hour
  minıimum=never maximum=always

CONTACTS AND LOCATIONS:
Overall Officials: GÜLCAN DÜRÜST SAKALLI, lecturer, Principal Investigator — Doğu Akdeniz Üniversitesi
Locations (3):
- Cyprus (3):
  - Gazimağusa Devlet Hastanesi (Eastern Mediterranean University), Famagusta, Northern Cyprus
  - Eastern Mediterranean University (Gazimağusa Devlet Hastanesi), Gazimağusa (Famagusta, North Cyprus), Northern Cyprus
  - Doğu Akdeniz Üniveristesi, Famagusta

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- See also: The effect of coffee/caffeine on postoperative ileus following elective colorectal surgery: a meta-analysis of randomized controlled trials — https://www.ncbi.nlm.nih.gov/pmc/articles/PMC8885519/
- See also: Effect of Coffee on the Length of Postoperative Ileus After Elective Laparoscopic Left-Sided Colectomy: A Randomized, Prospective Single-Center Study. — https://europepmc.org/article/MED/26445179
- See also: The Effect of Fennel Tea Drinking on Postoperative Gut Recovery after Gynecological Malignancies Operation — https://europepmc.org/article/MED/26867333